CLINICAL TRIAL: NCT07176923
Title: A Clinical Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of CS-121, an In Vivo Base Editing Therapy Delivered by Lipid Nanoparticles Targeting APOC3, in Adults With Familial Chylomicronemia Syndrome
Brief Title: CS-121 APOC3 Base Editing in FCS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CorrectSequence Therapeutics Co., Ltd (Industry)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS-121-01
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Familial Chylomicronemia Syndrome (FCS)
Keywords: Familial Chylomicronemia Syndrome (FCS); Severe Hypertriglyceridemia; Acute Pancreatitis; Apolipoprotein C3 (APOC3); In Vivo Base Editing; Lipid Nanoparticles (LNP); Gene Editing Therapy; First-in-Human Study; Rare Metabolic Disorder
MeSH Terms: conditions — Familial hyperchylomicronemia syndrome; Hypertriglyceridemia; Pancreatitis

STUDY DESIGN:
Intervention Model Description: About 3-15 participants with NAFCS ≥45 and fasting triglycerides ≥10 mmol/L will be enrolled. The study follows an adaptive design with three ascending dose levels and up to two de-escalation cohorts if needed. Each cohort includes 1-3 participants; escalation proceeds after ≥14 days of safety, PK, and PD review. A single intravenous infusion of CS-121 is given, followed by 5 days of inpatient monitoring and ~10 months of follow-up to assess safety, tolerability, PK, PD, and exploratory efficacy including triglyceride reduction and pancreatitis incidence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Single Low Dose CS-121 (Experimental): Participants in this arm will receive a single low dose of CS-121.
  Interventions: Biological: CS-121
- Single Middle Dose CS-121 (Experimental): Participants in this arm will receive a single middle dose of CS-121.
  Interventions: Biological: CS-121
- Single High Dose CS-121 (Experimental): Participants in this arm will receive a single high dose of CS-121.
  Interventions: Biological: CS-121
- Single Lower Dose 1 of CS-121 (Experimental): Participants in this arm will receive a single lower dose 1 of CS-121.
  Interventions: Biological: CS-121
- Single Lower Dose 2 of CS-121 (Experimental): Participants in this arm will receive a single lower dose 2 of CS-121.
  Interventions: Biological: CS-121

INTERVENTIONS:
Biological: CS-121 — CS-121 is a in vivo base editing therapy formulated in lipid nanoparticles for targeted editing of the APOC3 gene in hepatocytes. In this study, participants receive a single intravenous infusion of CS-121 at escalating dose levels. The investigational product is designed to reduce ApoC3 protein expression and serum triglyceride levels in adults with familial chylomicronemia syndrome (FCS).

SUMMARY:
This is an open-label, single-arm, dose-escalation Phase I clinical trial to evaluate the safety, tolerability, pharmacodynamics (PD), and pharmacokinetics (PK) of CS-121, an in vivo base editing therapy delivered by lipid nanoparticles targeting APOC3, in adult participants (18-55 years) with familial chylomicronemia syndrome (FCS).

DETAILED DESCRIPTION:
Familial chylomicronemia syndrome (FCS) is a rare, autosomal recessive lipid metabolism disorder characterized by impaired clearance of triglyceride-rich lipoproteins due to deficiencies in lipoprotein lipase or its cofactors. Patients experience severe hypertriglyceridemia, recurrent episodes of acute pancreatitis, abdominal pain, and other complications that significantly reduce quality of life and may be life-threatening. Despite strict dietary restrictions and conventional lipid-lowering therapies, many patients fail to achieve adequate triglyceride control, highlighting a major unmet medical need.

CS-121 is an investigational, in vivo base editing therapy delivered by lipid nanoparticles (LNPs) targeting the APOC3 gene in the liver. By introducing precise base edits at specific APOC3 loci, CS-121 is intended to mimic naturally occurring protective mutations that reduce ApoC3 expression, thereby restoring triglyceride clearance pathways and lowering pancreatitis risk. Preclinical studies in transgenic mouse and non-human primate models demonstrated dose-dependent APOC3 editing, reductions in serum ApoC3 protein and triglyceride levels, and acceptable safety profiles, supporting advancement into first-in-human evaluation.

This Phase I study uses an adaptive, dose-escalation design to investigate multiple dose levels of CS-121 in adults with genetically and clinically confirmed FCS. The design incorporates dynamic dose adjustment based on emerging safety, pharmacokinetic (PK), and pharmacodynamic (PD) data, consistent with regulatory guidance for rare disease trials.

Participants will undergo screening to confirm eligibility, including fasting triglyceride measurements, North American FCS score (NAFCS), genetic and laboratory testing, and imaging studies. Eligible participants will receive a single intravenous infusion of CS-121 and will be observed in-clinic immediately post-dose for early safety monitoring. Extended follow-up visits will be conducted for up to 10 months, with evaluations of clinical safety parameters, ApoC3 protein and triglyceride levels, drug exposure (sgRNA/mRNA), and exploratory endpoints such as pancreatitis incidence and imaging of hepatic lipid accumulation.

The study is designed to establish a dose range, identify an optimal biological dose (OBD), and provide first-in-human safety, tolerability, PK, and PD data for CS-121 in FCS. Findings from this trial will inform the future development of base editing therapies in severe hypertriglyceridemia and related rare metabolic disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years (inclusive) at the time of signing informed consent.
* On regular standard therapy with good compliance, but fasting triglyceride (TG) levels have not been consistently reduced below 10 mmol/L (880 mg/dL); i.e., before screening, there must be records of at least three separate fasting TG values >10 mmol/L (880 mg/dL), or the participant is intolerant to standard therapy.
* North American Familial Chylomicronemia Syndrome (NAFCS) score ≥45
* Able to sign informed consent and comply with the requirements and restrictions specified in the informed consent form and the protocol, such as dietary guidance and intake restrictions.
* Female participants must meet one of the following: be not of childbearing potential (e.g., documented hysterectomy, bilateral salpingectomy/sterilization, or ≥1 year postmenopausal); or, if of childbearing potential, have a negative pregnancy test at screening and be willing to use strict and effective contraception (e.g., abstinence, pharmacologic, or barrier methods) during the study. Male participants with reproductive potential must agree to use strict and effective contraception (e.g., abstinence, pharmacologic, or barrier methods) throughout the entire post-dose observation period; males without reproductive potential must provide supporting medical history (e.g., post-vasectomy).

Exclusion Criteria:

* Currently participating in another interventional clinical study, or last use of another investigational product with a washout period of less than 5 half-lives or 30 days (whichever is longer).
* Use of APOC3-targeted antisense oligonucleotides (ASO) or siRNA lipid-lowering agents within 6 months prior to dosing.
* History of acute pancreatitis within 3 months before dosing.
* History of acute coronary syndrome (ACS) within 6 months before dosing, such as myocardial infarction or unstable angina, or prior coronary revascularization (e.g., coronary artery bypass grafting, angioplasty, or stent implantation).
* In the investigator's judgment, receipt of major surgery within 3 months before dosing that would make the participant unsuitable for this study drug or unable to tolerate possible cytokine-release events.
* Any of the following laboratory abnormalities at screening:

ALT or AST ≥3 × ULN Total bilirubin ≥1.5 × ULN eGFR <30 mL/min/1.73 m² Random urine albumin-to-creatinine ratio (UACR) >30 mg/g LDL-C >130 mg/dL (3.4 mmol/L) HbA1c ≥9%

* Coagulation abnormalities deemed by the investigator to make CS-121 administration unsuitable.
* Positive at screening for HBsAg, HCV antibody and RNA, HIV, or Treponema pallidum (syphilis).
* Known major organ disease, psychiatric disorders, Cushing's syndrome, or malignancy that, in the investigator's judgment, would make the participant unsuitable for the study or unable to tolerate possible cytokine-release-like events.
* Concomitant medications or treatments judged by the investigator to affect lipid metabolism, hepatic or renal function, or coagulation, or to interfere with the evaluation of study drug efficacy, including but not limited to: systemic glucocorticoids, anabolic steroids, antiretroviral agents used within 4 weeks prior to dosing, plasma exchange, blood donation, or blood loss >200 mL.
* Planning pregnancy, currently pregnant, or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Events (TEAEs) | From the start of dosing through approximately 10 months of follow-up
  Incidence, nature, and severity of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs), adverse events of special interest (AESIs), and abnormalities in clinical symptoms, vital signs, physical examinations, laboratory tests, and electrocardiograms (ECGs). Severity will be graded according to NCI CTCAE version 5.0.
Dose-Limiting Toxicities (DLTs) | Number and type of dose-limiting toxicities (DLTs), defined as CTCAE grade ≥3 adverse events considered possibly, probably, or definitely related to CS-121 and persisting ≥7 days, or other adverse events/laboratory abnormalities that lead to suspension o
  Within 14 days after CS-121 infusion

SECONDARY OUTCOMES:
Change from Baseline in Fasting Serum Triglycerides (TG) | Baseline through approximately 10 months after dosing
  Absolute and relative change in fasting serum triglyceride levels compared with baseline values.
Change from Baseline in Serum ApoC3 Protein Levels | Baseline through approximately 10 months after dosing
  Absolute and relative change in serum ApoC3 protein concentrations compared with baseline values.
Peak Concentration (Cmax) of CS-121 Components | From dosing through approximately 1 month after infusion.
  Maximum observed concentration of CS-121 components following intravenous infusion.
Time to Maximum Concentration (Tmax) of CS-121 Components | From dosing through approximately 1 month after infusion
  Time to reach maximum observed concentration of CS-121 components following intravenous infusion
Area Under the Curve (AUC) of CS-121 Components | From dosing through approximately 1 month after infusion.
  Area under the Curve of CS-121 components to characterize systemic exposure

CONTACTS AND LOCATIONS:
Overall Officials: YALIANG LI, Study Director — CorrectSequence Therapeutics (Shanghai) Co., Ltd
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided